CLINICAL TRIAL: NCT05557981
Title: A Randomized Controlled Trial on The Impact of a Novel Coaching Program on Medical Errors, Clinical Reasoning, and Well-Being of Physicians, or the CARE (Coaching to Advance Resilience and Reduce Error) Study
Brief Title: The Impact of a Novel Coaching Program on Medical Errors and Well-Being of Physicians
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Harvard Risk Management Foundation (Other)
Responsible Party: Principal Investigator, Ritika S. Parris, Primary care physician, Director of Wellness for GME, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021P000482
Record Dates: First submitted 2022-09-22; First posted 2022-09-28 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Burnout; Adverse Event; Medical Education
Keywords: Coaching; burnout; wellness; medical errors
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Trainees - treatment (Experimental): Residents and fellows paired with a faculty coach from the "faculty - treatment" arm to participate in up to 4 coaching meetings
  Interventions: Behavioral: Coaching
- Trainees - control (No Intervention): Residents and fellows randomized to the control arm. They are not paired with a faculty coach and instead continue to receive standard mentorship as part of their training program.
- Faculty - treatment (Experimental): Faculty members randomized to receive coaching training and are paired with a resident/fellow from the "trainees - treatment" arm to conduct up to 4 coaching sessions over the course of the academic year.
  Interventions: Behavioral: Coaching
- Faculty - control (No Intervention): Faculty members randomized to control arm. They are not paired with a trainee from this study and instead continue to provide mentorship as they typically would, as part of their role at an academic medical center

INTERVENTIONS:
Behavioral: Coaching — A novel coaching curriculum based in positive psychology with an emphasis on self-reflection, goal setting and adverse event processing.
  Arms: Faculty - treatment; Trainees - treatment

SUMMARY:
This is a randomized controlled trial with a mixed method design to determine the impact of coaching on self-perceived medical errors, burnout, and resilience. The study team developed a novel coaching curriculum based in principles of positive psychology and self-reflection with the hypothesis that the coaching intervention will lead to decreased medical errors, decreased burnout, and increased resilience in trainee and faculty participants. Resident and fellow trainees as well as faculty members were recruited across departments and randomized to coaching or control. Faculty in the coaching arm were trained in coaching techniques and paired with a trainee coachee. Survey results as well as focus groups will be used to analyze the impact of the coaching program as compared to standard mentorship (control).

ELIGIBILITY:
Inclusion Criteria:

* Residents and fellows in a training program at Beth Israel Deaconess Medical Center (BIDMC)
* faculty members at BIDMC

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Medical errors in trainees | baseline (pre) compared to results at the end (post) of the coaching intervention, an average of 9 months
  Self-perceived medical errors amongst trainees based on survey response.
Burnout | baseline (pre) compared to results at the end (post) of the coaching intervention, an average of 9 months
  Burnout score amongst trainees and faculty based on Stanford Professional Fulfillment Index
Resilience | baseline (pre) compared to results at the end (post) of the coaching intervention, an average of 9 months
  Burnout score amongst trainees and faculty based on Connor Davidson Resilience Scale 2

SECONDARY OUTCOMES:
medical errors in faculty | baseline (pre) compared to results at the end (post) of the coaching intervention, an average of 9 months
  Self-perceived medical errors amongst faculty based on survey response. Specifically, faculty are asked "Do you think you may have made any medical error in the last 3 months? A medical error is the failure of a planned action to be completed as intended, or the failure of an unplanned action that should have been completed" with answer choices yes, no, and unsure.
delayed medical errors in faculty | baseline (beginning of study, before intervention) compared to 6 months post coaching program
  Self-perceived medical errors amongst faculty based on survey response
Mechanism of change | assessed an average of 1 year after intervention initiation
  Mechanism of change in burnout, resilience and medical errors in both trainees and faculty as compared to standard mentorship
Delayed Medical errors in trainees | up to 15 months
  Self-perceived medical errors amongst trainees based on survey response
Burnout | baseline (beginning of study, before intervention) compared to 6 months post coaching program
  Burnout score amongst trainees and faculty based on Stanford Professional Fulfillment Index
Delayed Resilience | baseline (beginning of study, before intervention) compared to 6 months post coaching program
  Burnout score amongst trainees and faculty based on Connor-Davidson-RISC2

CONTACTS AND LOCATIONS:
Overall Officials: Ritika Parris, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States